CLINICAL TRIAL: NCT05370092
Title: Effect of Percutaneous Needle Electrolysis on Tibialis Posterior Tendinopathy
Brief Title: Effect of Percutaneous Needle Electrolysis (PNE) on Tendinopathy
Acronym: PNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Antonio Rejas Fenández, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1801202201622
Record Dates: First submitted 2022-03-31; First posted 2022-05-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Posterior Tibial Tendon Dysfunction
MeSH Terms: conditions — Posterior Tibial Tendon Dysfunction | interventions — Exercise Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients assigned to this group will receive a session of manual therapy and therapeutic exercise. The manual therapy (TM) treatment for tendinopathies is mainly focused on soft tissue mobilization and deep transverse friction massage (Cyriax).
  The therapeutic exercise session participants will perform 2 exercises for 4 weeks 3 days per week. The first exercise they will perform will be the Short-Foot Exercise holding the position 5 seconds isometrically. The second exercise will be plantar flexion of the ankle with adduction of the foot and inversion with elastic band in its concentric and eccentric phase. Each exercise will be performed in 3 series of 15 repetitions, with 1 minute rest between series, the exercise session will follow the TM and will last approximately 15-20 minutes.
  Interventions: Other: Therapeutic exercise; Other: Manual therapy
- Intervention group (Experimental): Participants in this group will receive 4 sessions (once a week during their respective treatment session) of percutaneous electrolysis guided by MUSCULO-SKELETAL ECOGRAPHY, by a physiotherapist with extensive clinical experience in this therapeutic approach. The technique will be applied using a specifically developed and medically certified device (EPI Advanced Medicine®, Barcelona, Spain. EPI®). The galvanic current will be applied using acupuncture needles. In the present study, a 0.30*25 mm needle (Agupunt, Barcelona, Spain) will be used, with an intensity of 2 mA for a total of 3-5 seconds and 3-5 impacts on the liquid content (TTP tenosynovitis) and 2 mA for a total of 3 seconds and 2-3 impacts if in the tendon (intrasubstance). The technique shall be applied under ultrasound guidance.
  The needle shall be introduced at an angle of 80° in a short-axis cross-section to the skin, with the tip of the needle directed towards the posterior tibial tendon.
  Interventions: Other: Percutaneous needle electrolysis; Other: Therapeutic exercise; Other: Manual therapy

INTERVENTIONS:
Other: Percutaneous needle electrolysis — Electrolysis is the process by which water (H2O) and sodium chloride (NaCl) molecules, which are present in the biological tissues and body compartments of our organism, are organically broken down into their constituent chemical elements, regrouping to create entirely new substances such as sodium hydroxide (NaOH), hydrogen gas (H2) and chlorine gas (Cl2). This process occurs thanks to the passage of a flow of direct electric current, also known as galvanic current, which is a totally athermal process. The passage of this current allows a local inflammatory response to occur (increase in lymphocytes and macrophages) as well as an increase in vasodilatation, inducing phagocytosis and biological stimulation of tendon repair.
  Arms: Intervention group
Other: Therapeutic exercise — The first exercise they will perform will be the Short-Foot Exercise holding the position 5 seconds isometrically. The second exercise will be plantar flexion of the ankle with adduction of the foot and inversion with elastic band in its concentric and eccentric phase
Other: Manual therapy — The manual therapy (TM) treatment for tendinopathies is mainly focused on soft tissue mobilization and deep transverse friction massage (Cyriax).

SUMMARY:
The aim of this study is to test the efficacy of percutaneous electrolysis in posterior tibial tendinopathies. The posterior tibial tendon injury is one of the most frequent pathologies in the lower extremities, and therefore a correct study and evaluation of it is necessary. This study aims to compare the therapeutic effect of percutaneous electrolysis comparing a control group with an experimental group. To evaluate functionality, pain and its ultrasound pattern before and after treatment, in order to assess the efficacy of the treatment.

DETAILED DESCRIPTION:
A single-blind, longitudinal, randomised, controlled, single-blind, longitudinal, randomised, controlled clinical trial will be conducted. First, the participant will receive a FOOT AND ANKLE ABILITY (FAAM) survey, along with a numerical pain scale, both of which must be completed. Next, an ultrasound study of the foot will be performed, focusing on pain in the inner ankle, to check for possible pathology in the posterior tibial tendon. Finally, the physiotherapist's intervention will be carried out to check the effectiveness of the technique, which may cause some pain, and finally, the numerical pain scale will be passed again. Four sessions will be carried out in four different weeks, always using the same day of the week for the intervention and following the same steps as above. The purpose of this study is to test the efficacy of PD in posterior tibial tendinopathy and whether PD is therefore a safe technique for this type of intervention. All patients will sign an informed consent form and will be informed about the study beforehand.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age
* Mild inflammation, swelling and/or tenderness posterior to the medial malleolus
* Pain posterior and/or superior to the medial malleolus, aggravated by activity
* Pain present for at least 3 months
* One or more signs of flexible flatfoot deformity, including excessive valgus deformity of the hindfoot during weight bearing and/or excessive foot abduction (many toes sign).
* Pain when performing the Hell Rise Test or performed incorrectly.
* Signs of tenosynovitis on ultrasound examination.

As the inclusion criteria are based on side-to-side comparison all participants had to have unilateral involvement.

Exclusion Criteria:

* Previous surgery on the affected foot, leg or knee.
* Disabling osteoarthritis of the knee on the affected side.
* Fixed hindfoot deformities.
* Recurrent ankle sprains on the affected side.
* Ligament tears or bony abnormalities of the affected foot.
* A physical or medical condition that contraindicates the testing protocol.
* Pregnancy.
* FCD or FLH tendinopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
NUMERICAL PAIN RATE SCALE (NPRS. 0-10) | 6 months
  The scale consists of a horizontal line of 11 numbers, at the ends of which are the extreme manifestations of a symptom that allows observers to measure the intensity of pain with maximum reproducibility. On the far left is 0 or the total absence of pain and on the far right is 10 or the maximum pain that can be tolerated. The patient will be asked to select the number where they consider their pain to be.

SECONDARY OUTCOMES:
FOOT AND ANKLE ABILITY (FAAM) | 6 months
  The FAAM questionnaire consists of 29 items separated into two subscales: the ADL subscale with 21 items and the Sport subscale with 8 items. Each one has a maximum Likert scale score of 5 points ranging from "no difficulty" to "impossible to perform". All scores will be converted to percentages, with a higher percentage indicating a higher level of functionality and lower pathology. At the end of the scale, the functionality percentage will be calculated, ranging from 0% (inability to perform any activity) to 100% (normal functionality level). Finally, patients will rate the condition of their ankle and foot on a 4-point scale that includes "normal," "almost normal," "abnormal," and "severely abnormal." The intention of the study is that the patient recovers 100% of functionality or better the percentage that has been marked prior to the intervention. As in the 4-point scale, the condition of your ankle should be normal.

OTHER OUTCOMES:
ULTRASOUND CONTROL | 4 weeks
  All participants, both in the control and experimental groups, will be examined before the intervention and at the end of the 4 sessions to evaluate possible changes in the tendon, and all invasive interventions will be performed ultrasonographically. This measurement was just a qualitative control of the diagnosis of tendinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Rejas Fernández, Principal Investigator — Universidad Rey Juan Carlos; Jose Luis Arias Buría, Study Director — Universidad Rey Juan Carlos; Ana Isabel De La Llave Rincón, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abat F, Gelber PE, Polidori F, Monllau JC, Sanchez-Ibanez JM. Clinical results after ultrasound-guided intratissue percutaneous electrolysis (EPI(R)) and eccentric exercise in the treatment of patellar tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2015 Apr;23(4):1046-52. doi: 10.1007/s00167-014-2855-2. Epub 2014 Jan 30. PMID 24477495
- [Background] Abat F, Diesel WJ, Gelber PE, Polidori F, Monllau JC, Sanchez-Ibanez JM. Effectiveness of the Intratissue Percutaneous Electrolysis (EPI(R)) technique and isoinertial eccentric exercise in the treatment of patellar tendinopathy at two years follow-up. Muscles Ligaments Tendons J. 2014 Jul 14;4(2):188-93. eCollection 2014 Apr. PMID 25332934
- [Background] Margalef R, Bosque M, Minaya-Munoz F, Valera-Garrido F, Santafe MM. Safety analysis of percutaneous needle electrolysis: a study of needle composition, morphology, and electrical resistance. Acupunct Med. 2021 Oct;39(5):471-477. doi: 10.1177/0964528420988007. Epub 2021 Feb 7. PMID 33550820
- [Background] Lopez-Royo MP, Gomez-Trullen EM, Ortiz-Lucas M, Galan-Diaz RM, Bataller-Cervero AV, Al-Boloushi Z, Hamam-Alcober Y, Herrero P. Comparative study of treatment interventions for patellar tendinopathy: a protocol for a randomised controlled trial. BMJ Open. 2020 Feb 16;10(2):e034304. doi: 10.1136/bmjopen-2019-034304. PMID 32066608
- [Background] Arias-Buria JL, Truyols-Dominguez S, Valero-Alcaide R, Salom-Moreno J, Atin-Arratibel MA, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrolysis and Eccentric Exercises for Subacromial Pain Syndrome: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:315219. doi: 10.1155/2015/315219. Epub 2015 Nov 15. PMID 26649058
- [Background] Gomez-Chiguano GF, Navarro-Santana MJ, Cleland JA, Arias-Buria JL, Fernandez-de-Las-Penas C, Ortega-Santiago R, Plaza-Manzano G. Effectiveness of Ultrasound-Guided Percutaneous Electrolysis for Musculoskeletal Pain: A Systematic Review and Meta-Analysis. Pain Med. 2021 May 21;22(5):1055-1071. doi: 10.1093/pm/pnaa342. PMID 33155055
- [Background] Cook JL, Purdam CR. Is tendon pathology a continuum? A pathology model to explain the clinical presentation of load-induced tendinopathy. Br J Sports Med. 2009 Jun;43(6):409-16. doi: 10.1136/bjsm.2008.051193. Epub 2008 Sep 23. PMID 18812414
- [Background] Rabbito M, Pohl MB, Humble N, Ferber R. Biomechanical and clinical factors related to stage I posterior tibial tendon dysfunction. J Orthop Sports Phys Ther. 2011 Oct;41(10):776-84. doi: 10.2519/jospt.2011.3545. Epub 2011 Jul 12. PMID 21765219
- [Background] Johnson KA, Strom DE. Tibialis posterior tendon dysfunction. Clin Orthop Relat Res. 1989 Feb;(239):196-206. PMID 2912622
- [Background] Mills FB 4th, Williams K, Chu CH, Bornemann P, Jackson JB 3rd. Prevalence of Abnormal Ultrasound Findings in Asymptomatic Posterior Tibial Tendons. Foot Ankle Int. 2020 Sep;41(9):1049-1055. doi: 10.1177/1071100720931085. Epub 2020 Jun 21. PMID 32567358
- [Background] Bellew SD, Colbenson KM, Bellamkonda VR. Posterior Tibial Tendon Tenosynovitis Diagnosed by Point-of-Care Ultrasound. Clin Pract Cases Emerg Med. 2017 Oct 18;1(4):439-440. doi: 10.5811/cpcem.2017.6.34430. eCollection 2017 Nov. No abstract available. PMID 29849380
- [Background] Ikpeze TC, Brodell JD Jr, Chen RE, Oh I. Evaluation and Treatment of Posterior Tibialis Tendon Insufficiency in the Elderly Patients. Geriatr Orthop Surg Rehabil. 2019 Jan 24;10:2151459318821461. doi: 10.1177/2151459318821461. eCollection 2019. PMID 30719400
- [Background] Ross MH, Smith MD, Mellor R, Vicenzino B. Exercise for posterior tibial tendon dysfunction: a systematic review of randomised clinical trials and clinical guidelines. BMJ Open Sport Exerc Med. 2018 Sep 19;4(1):e000430. doi: 10.1136/bmjsem-2018-000430. eCollection 2018. PMID 30271611
- [Background] Sanchez-Sanchez JL, Calderon-Diez L, Herrero-Turrion J, Mendez-Sanchez R, Arias-Buria JL, Fernandez-de-Las-Penas C. Changes in Gene Expression Associated with Collagen Regeneration and Remodeling of Extracellular Matrix after Percutaneous Electrolysis on Collagenase-Induced Achilles Tendinopathy in an Experimental Animal Model: A Pilot Study. J Clin Med. 2020 Oct 15;9(10):3316. doi: 10.3390/jcm9103316. PMID 33076550
- [Background] Millar NL, Silbernagel KG, Thorborg K, Kirwan PD, Galatz LM, Abrams GD, Murrell GAC, McInnes IB, Rodeo SA. Tendinopathy. Nat Rev Dis Primers. 2021 Jan 7;7(1):1. doi: 10.1038/s41572-020-00234-1. PMID 33414454